CLINICAL TRIAL: NCT02656979
Title: Blood Flow of Ophthalmic Artery and Its Relationship to Structural Properties of the Optic Nerve and Intraocular Pressure in Glaucoma
Brief Title: Blood Flow of Ophthalmic Artery and Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UmeaU
Record Dates: First submitted 2015-12-15; First posted 2016-01-15 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Blood flow; Pseudoexfoliation; Intraocular pressure; Brain perfusion; Magnetic Resonance Imaging
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood flow pre&post IOP lowering (Other): After measurement of blood flow with MRI and measurements of ocular parameters the patient receives the IOP lowering eye drop latanoprost once daily in one eye for approximately one week and then the measurements are are repeated in the same manner.
  Interventions: Drug: Latanoprost
- Blood flow (No Intervention): The subjects will do blood flow measurements with MRI and measurements of ocular parameters only once. No intervention with IOP lowering drops.

INTERVENTIONS:
Drug: Latanoprost — Between measurements on day 1 and day 2, the subjects will receive a drop of latanoprost which is an IOP lowering drug once daily in one eye.
  Arms: Blood flow pre&post IOP lowering

SUMMARY:
The main purpose of this project is to investigate the blood flow of the ophthalmic artery (OA) in patients with ocular hypertension, high tension glaucoma and normal tension glaucoma. It is also to study the influence of the intraocular pressure difference on OA blood flow in the two first groups. Furthermore, the investigators want to understand the relationship between ocular dynamics, blood flow and structural alternations of the optic nerve head (ONH). The rationale behind the study is to improve knowledge of the pathogenesis of glaucoma.

DETAILED DESCRIPTION:
The investigators will investigate the OA blood flow, intraocular pressure (IOP) and structural properties of the optic nerve. The investigators will include glaucoma patients as they believe that glaucoma may be caused by or influenced by OA blood flow. The investigators will include also patients with intraocular hypertension with and without pseudoexfoliation in order to study how changes in IOP interact with OA blood flow and the structural properties of the optic nerve in a group that does not develop glaucoma. In addition, the investigators will investigate patients that develop glaucoma in spite of a normal IOP. Therefore, the investigators will study three fundamentally different groups (G1, G2 and G3) of patients as well as a control group of healthy subjects (G4):

G1: Newly diagnosed and untreated Glaucoma (optic and visual field damage exists).

G2: Ocular hypertension with IOP ≥ 23 mmHg (i.e. only elevated eye pressure).

G3: Normal Tension Glaucoma.

G4: Healthy subjects.

Each group will include 25 patients apart from G2 where 50 patients will be included, half of which have pseudoexfoliation syndrome. The study will be performed in accordance with the tenets of the Helsinki Declaration and is approved by the regional ethical board.

Study protocol overview:

Study protocol consists of two parts of examinations repeated with approximately one week between: Each part is divided into two examinations; one at the Department of radiology followed by one at the Department of ophthalmology. The measurements are repeated approximately one week later for G1 and G2.

Day 1: First, MRI scans on the brain to measure the blood flow of OA as well as the structural and morphological properties of the ON (see method below). Second, just after MRI examination, the patient will be examined at the Department of ophthalmology. Measurement of intraocular pressure, ocular pulse amplitude, central corneal thickness, bulb length, investigation with optical coherence tomography (OCT) and blood pressure will be performed. The patients from G3 (Normal Pressure Glaucoma) will participate only in Day 1, since most cases already has pressure-lowering treatment. Also subjects in G4 vill only participate in Day 1. All other participants will receive pressure lowering drug (Latanoprost) in one eye once daily, until the protocol is repeated at Day 2.

Day 2: The measurements at Day 1 are repeated approximately one week later. The measurements will be made in both eyes, which is why an eye can serve as a control. That way the investigators will have a good opportunity to assess how much of the change the investigators see in the treated eye that may be due to normal variations in OA blood flow and how much depends on the given treatment.

The findings will be compared between the groups and to the normal material in G4. The investigators will be able to see whether, and if so, to what extent, eyes with glaucoma differ from normal eyes in terms of blood flow through OA as compared to the IOP measurements, and different biomechanical parameters of the eye. Thus, determine the pressure dynamics and calculate ocular compliance with the three different groups of research subjects; newly diagnosed glaucoma, ocular hypertension, normal tension glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and untreated glaucoma patients
* Treated normal tension glaucoma patients
* Untreated patients with ocular hypertension
* Subjects with healthy eyes

Exclusion Criteria:

* Heart disease except treated hypertension
* Intracranial pathology such as stroke, tumor, previous intracranial surgery
* Insulin treated diabetes mellitus

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2013-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The blood flow (ml/min) of the ophthalmic artery in patients with different types of glaucoma/ocular hypertension and healthy individuals will be measured with MRI | Up to four years

SECONDARY OUTCOMES:
The change of ophthalmic artery blood flow (ml/min) after a reduction in IOP in glaucoma and intraocular hypertension will be measured with MRI | Up to four years
The change of structural properties (μm) of the optic nerve after a reduction in IOP in glaucoma and intraocular hypertension will be measured with MRI | Up to four years
Difference in the ophthalmic artery blood flow (ml/min) measured with MRI in patients with ocular hypertension with and without pseudoexfoliation. | Up to four years

CONTACTS AND LOCATIONS:
Overall Officials: Gauti Jóhannesson, M.D., Ph.D., Principal Investigator — Department of Clinical Science, Ophthalmology, Umeå University
Locations (1):
- Department of Clinical Science, Ophthalmology, Umeå University, Umeå, Västerbotten County, Sweden